CLINICAL TRIAL: NCT00428623
Title: Aquacel Compared to Traditional Post Surgical Wound Dressing in Vascular Surgery Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: Torben V Schroeder
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Wound Healing; Patient Comfort
Keywords: Patient comfort; Wound dressings; infection; vascular surgery
MeSH Terms: conditions — Infections | interventions — Bandages

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: wound dressing

SUMMARY:
The study is a prospective randomised, controlled study of 136 patients undergoing vascular surgery. Their closed wounds were covered with either aquacel, a hydrofiber dressing, or a traditional gauze dressing.Number of changes, patient comfort,number of infections, length of hospital stay and wound complications were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective vascular surgery, with an expected hospital stay of at least 4 days. informed consent

Exclusion Criteria:

* known hypersensitivity to the dressing materials. age under 18 years. dementia, insufficient danish language understanding, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-01; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: torben V Schroeder, prof,dmsc.md, Study Director — professor
Locations (1):
- Department of Vascular Surgery, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835